CLINICAL TRIAL: NCT03146793
Title: National Follow-up of Dialysis Patients With Sodium Thiosufate-treated Calciphylaxis Under Temporary Use Authorization
Brief Title: The Early Administration of Sodium Thiosulfate Should Help to Reduce the Mortality of Dialysis Patients With Calciphylaxis, From a National Cohort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier St Esprit (Other)
Responsible Party: Principal Investigator, Albert TRINH-DUC, Principal investigator, Centre Hospitalier St Esprit
Other Study IDs: Centre Hospitalier St Esprit
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Calciphylaxis; Renal Insufficiency, Chronic
Keywords: Calciphylaxis/complications; Kidney Failure, Chronic/complications; Renal Dialysis; Thiosulfates/therapeutic use; Time Factors
MeSH Terms: conditions — Calciphylaxis; Renal Insufficiency, Chronic; Renal Insufficiency; Bronchiolitis Obliterans Syndrome | interventions — sodium thiosulfate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Sodium Thiosulfate — 25g intravenously 3 times per week

SUMMARY:
The national drug safety agency authorizes nominatively the use of sodium thiosulfate in dialysis patients with calciphylaxis. To date, it is the largest global cohort (more 600 patients from 2012 to 2016). We wanted to study retrospectively the fate of these patients at 6 months including mortality. Early use improves effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* All dialysis patients with calciphylaxis in France who have obtained a temporary use authorization for sodium thiosulfate by National Agency for the Safety of Medicines

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dialysis patients with calciphylaxis
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-02-28 (Estimated)

PRIMARY OUTCOMES:
Mortality | 6 months

SECONDARY OUTCOMES:
time factor on mortality | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Albert TRINH-DUC, MD, Principal Investigator — Centre Hospitalier St EPSRIT AGEN FRANCE
Locations (1):
- Centre Hospitalier St ESPRIT, Agen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weenig RH, Sewell LD, Davis MD, McCarthy JT, Pittelkow MR. Calciphylaxis: natural history, risk factor analysis, and outcome. J Am Acad Dermatol. 2007 Apr;56(4):569-79. doi: 10.1016/j.jaad.2006.08.065. Epub 2006 Dec 1. PMID 17141359
- [Background] Perceau G. [Uraemic and non-uraemic calcific arteriopathy: The need for rapid diagnosis and therapy]. Ann Dermatol Venereol. 2015 Aug-Sep;142(8-9):506-12. doi: 10.1016/j.annder.2015.06.009. Epub 2015 Aug 5. French. PMID 26253008
- [Background] Nigwekar SU, Brunelli SM, Meade D, Wang W, Hymes J, Lacson E Jr. Sodium thiosulfate therapy for calcific uremic arteriolopathy. Clin J Am Soc Nephrol. 2013 Jul;8(7):1162-70. doi: 10.2215/CJN.09880912. Epub 2013 Mar 21. PMID 23520041
- [Background] Brandenburg VM, Kramann R, Rothe H, Kaesler N, Korbiel J, Specht P, Schmitz S, Kruger T, Floege J, Ketteler M. Calcific uraemic arteriolopathy (calciphylaxis): data from a large nationwide registry. Nephrol Dial Transplant. 2017 Jan 1;32(1):126-132. doi: 10.1093/ndt/gfv438. PMID 26908770
- [Background] Sood AR, Wazny LD, Raymond CB, Leung K, Komenda P, Reslerova M, Verrelli M, Rigatto C, Sood MM. Sodium thiosulfate-based treatment in calcific uremic arteriolopathy: a consecutive case series. Clin Nephrol. 2011 Jan;75(1):8-15. PMID 21176746